CLINICAL TRIAL: NCT06027801
Title: Iron Fortified Food to Improve Japanese Encephalitis and Typhoid Fever Vaccine Immunogenicity: a Randomized Controlled Trial in Iron Deficient Thai Women
Brief Title: Iron Fortified Food to Improve Japanese Encephalitis and Typhoid Fever Vaccine Immunogenicity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VEST
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-08

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron fortification group (Experimental): Participants assigned to this group will receive iron-fortified cookies daily for the whole study duration
  Interventions: Other: Iron-fortified cookies; Biological: Japanese encephalitis (JE) vaccine; Biological: Typhoid Vi polysaccharide (Vi-PS) vaccine
- Control group (Placebo Comparator): Participants assigned to this group will receive the same cookies containing no iron daily for the whole study duration
  Interventions: Biological: Japanese encephalitis (JE) vaccine; Biological: Typhoid Vi polysaccharide (Vi-PS) vaccine; Other: non-fortified cookies

INTERVENTIONS:
Other: Iron-fortified cookies — Study cookies fortified with ferrous fumarate, providing 15 mg of elemental iron in each portion.
  Arms: Iron fortification group
Biological: Japanese encephalitis (JE) vaccine — All participants will be administered the live attenuated JE vaccine
Biological: Typhoid Vi polysaccharide (Vi-PS) vaccine — All participants will be administered the typhoid Vi-PS vaccine
Other: non-fortified cookies — Study cookies containing no iron
  Arms: Control group

SUMMARY:
Iron deficiency (ID) anaemia (IDA) is a global public health problem, with the highest prevalence in Africa and in South-East Asia. While immunization programs have achieved high global coverage, vaccines often underperform in low- and middle-income countries (LMIC). The cause remains uncertain, but undernutrition, including ID, likely plays a role. Our recent in vitro and in vivo studies have shown the importance of iron status in adaptive immunity and vaccine response. Hypoferremia blunted T cell, B cell, and neutralizing antibody responses to influenza virus infection in mice, allowing the virus to persist. Iron deficient anaemic Kenyan women receiving intravenous iron at time of vaccination had a better immune response to the first dose of the ChAdOx Coronavirus 19 (COVID-19) vaccine and yellow fever vaccine. Japanese encephalitis and typhoid fever are endemic in Thailand. Vaccines are available but show variable efficacy. Whether ID impairs adult vaccine response to the live attenuated Japanese encephalitis (JE) and the Typhoid Vi polysaccharide (Vi-PS) vaccine and whether iron repletion via iron fortification improves vaccine response is uncertain.

The objective of this study is to assess whether IDA in Thai women impairs immune response to the JE and the Typhoid Vi-PS vaccine and whether fortification iron improves their response.

In this double-blind randomized controlled trial, IDA women will be assigned to two study groups: group 1 (fortification group) will receive iron-fortified biscuits (15mg iron as ferrous fumarate) for 56 days; group 2 (control group) will receive non-fortified biscuits for 56 days. All women will receive live attenuated JE and Typhoid Vi-PS vaccine on study day 28. Vaccine response will be measured 28 days after vaccination (on day 56) in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Female aged 18-49 years.
* Diagnosed with anaemia (i.e. hemoglobin (Hb) concentration <12 g/dl), but no severe anaemia (Hb <8 g/dl), and iron deficiency (ZnPP >40 µmol/mol)
* Anticipated residence in the area for the study duration

Exclusion Criteria:

* Pregnant (confirmed by rapid test during screening and at time of vaccination), lactating or planning pregnancy during the trial.
* Blood transfusion or intravenous iron treatment within 4 months of study start
* Major chronic infectious disease (e.g., tuberculosis, HIV+, hepatitis)
* Major chronic non-infectious disease (e.g., Type 1 or 2 diabetes, cancer)
* Treatment with supplemental iron two weeks prior to enrolment
* JE or typhoid vaccine within the past two years

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Immunoglobulin G (IgG) concentrations against Salmonella Typhi | day 28 (time of vaccination)
Immunoglobulin A (IgA) concentrations against Salmonella Typhi | day 28 (time of vaccination)
Immunoglobulin G (IgG) concentrations against Salmonella Typhi | day 56 (4 weeks after vaccination)
Immunoglobulin A (IgA) concentrations against Salmonella Typhi | day 56 (4 weeks after vaccination)
Neutralizing antibodies against Japanese encephalitis | day 28 (time of vaccination)
Neutralizing antibodies against Japanese encephalitis | day 56 (4 weeks after vaccination)

SECONDARY OUTCOMES:
Hemoglobin concentration (g/dL) | day 0
Hemoglobin concentration (g/dL) | day 28
Hemoglobin concentration (g/dL) | day 56
zinc protoporphyrin (ZnPP) concentration (µmol/mol heme) | day 0
zinc protoporphyrin (ZnPP) concentration (µmol/mol heme) | day 28
zinc protoporphyrin (ZnPP) concentration (µmol/mol heme) | day 56
serum iron (SFe) concentration (ng/µl) | day 0
serum iron (SFe) concentration (ng/µl) | day 28
serum iron (SFe) concentration (ng/µl) | day 56
total iron binding capacity (µg/dL) | day 0
total iron binding capacity (µg/dL) | day 28
total iron binding capacity (µg/dL) | day 56
transferrin saturation (TSAT) (%) | day 0
transferrin saturation (TSAT) (%) | day 28
transferrin saturation (TSAT) (%) | day 56
plasma ferritin (PF) concentration (µg/L) | day 0
plasma ferritin (PF) concentration (µg/L) | day 28
plasma ferritin (PF) concentration (µg/L) | day 56
soluble transferrin receptor (sTfR) concentration (mg/L) | day 0
soluble transferrin receptor (sTfR) concentration (mg/L) | day 28
soluble transferrin receptor (sTfR) concentration (mg/L) | day 56
C-reactive protein (CRP) concentration (mg/L) | day 0
C-reactive protein (CRP) concentration (mg/L) | day 28
C-reactive protein (CRP) concentration (mg/L) | day 56
alpha-glycoprotein (AGP) concentration (g/L) | day 0
alpha-glycoprotein (AGP) concentration (g/L) | day 28
alpha-glycoprotein (AGP) concentration (g/L) | day 56
retinol-binding protein concentration (µmol/L) | day 0
retinol-binding protein concentration (µmol/L) | day 28
retinol-binding protein concentration (µmol/L) | day 56

CONTACTS AND LOCATIONS:
Locations (1):
- Mahidol University, Roi Et, Thailand

IPD SHARING:
Plan to Share IPD: No